CLINICAL TRIAL: NCT01168102
Title: Noninvasive Blood Ethanol Measurement With Infrared Spectroscopy
Status: Completed | Type: Observational
Sponsor: InLight Solutions (Industry)
Collaborators: TruTouch Technologies (Unknown)
Responsible Party: Jeff Way, InLight Solutions
Other Study IDs: ILS-07-051
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2008-02

CONDITIONS: Healthy Individuals; At Least 21 Years of Age

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The objective of this study is to assess the performance of a noninvasive device for the detection of blood alcohol levels.

DETAILED DESCRIPTION:
The use and abuse of alcohol in the workplace, on our highways, and in public places is a significant national problem that affects and puts at risk almost all Americans. Alcohol-related accidents, crimes, and incidents continue to rise in the United States and across the world. Each year, alcohol-associated fatalities, injuries, and property losses cost our nation billions of dollars in medical and insurance costs, lost wages and productivity. Current technology for detecting and screening alcohol use and impairment, both at the workplace and while operating a vehicle, raises a number of concerns related to its accuracy, ease of use, and reliability in the field. This technology offers a low-cost, non-invasive method by which to measure blood alcohol. The device does not rely on human fluids and is coupled with the ability to verify identity. This will be greatly preferable to current standards, which require lengthy procedures and costly disposables.

InLight Solutions and TruTouch Technologies are developing a compact, robust alcohol sensor derived from a miniature home glucose meter. Initial conceptual testing, using synthetic data, demonstrates a system with better than 0.01% BAC error without requiring costly disposables or exposing the test administrator to any biohazards. The system offers the potential for untrained or minimally trained operators to achieve clinically and legally accurate measurements in less than 30 seconds. Additionally, an autonomous instrument could be configured to allow identification and monitoring of alcohol offenders without any further judicial involvement.

InLight Solutions technology employs advanced optical tissue sampling techniques and sophisticated multivariate analysis techniques (also known as "chemometrics") for quantitative near-infrared spectroscopy. These optical measurement techniques employ the painless use of light directed through human tissue to measure the chemical constituency of blood and tissue. These techniques can measure a variety of blood analytes, including alcohol.

An additional capability of the device is to be able to identify subjects based upon their unique skin spectra. This capability could be used when the technology is used as an ignition interlock device. Currently, a breath alcohol detection device is used to start an ignition interlock. This poses a problem due to the fact that users are able to have a different "sober" person blow into the device. Our technology could bypass this problem by using the device to both identify the user and their current blood alcohol level.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 21 but under the age of 70
2. No history of alcoholism -

Exclusion Criteria:

1. Pregnancy (Determined by Sure-Vue urine pregnancy test).
2. Females that have given birth within 1 month prior or are currently breastfeeding.
3. History of Alcoholism (Determined by MAST Test).
4. Under the age of 21 (All Subjects will have ID Checked).
5. Diagnosed with Type I or II Diabetes (Self-Reported). -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1. Over the age of 21 but under the age of 70
  2. No history of alcoholism -
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rohrscheib, M.D., Principal Investigator — UNMHSC
Locations (1):
- InLight Solutions, Albuquerque, New Mexico, United States

REFERENCES:
- See also: Related Info — http://www.inlightsolutions.com